CLINICAL TRIAL: NCT04109742
Title: Curcumin for Pediatric Nonalcoholic Fatty Liver Disease: A Pilot Randomized Controlled Trial
Brief Title: Curcumin for Pediatric Nonalcoholic Fatty Liver Disease
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Columbia University (Other)
Collaborators: Thorne HealthTech, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AAAS6731
Record Dates: First submitted 2019-09-23; First posted 2019-09-30 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: NAFLD - Nonalcoholic Fatty Liver Disease; NASH - Nonalcoholic Steatohepatitis
Keywords: Pediatric; NAFLD - nonalcoholic fatty liver disease; Curcumin; Fatty liver
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fatty Liver

STUDY DESIGN:
Intervention Model Description: The comparison of two different doses (500mg/qd and 1g/qd) of a phosphatidylcholine-curcumin complex supplement, to matching placebo
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participants, investigators, clinical staff, and data monitoring committee will not have knowledge of the interventions assigned to individual participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Curcumin 500mg capsules (Active Comparator): Dose will be 500mg daily phosphatidylcholine-curcumin complex supplement, orally for 24 weeks
  Interventions: Drug: phosphatidylcholine-curcumin complex supplement
- Curcumin 1000mg capsules (Active Comparator): Dose will be1g daily of phosphatidylcholine-curcumin complex supplement, orally for 24 weeks
  Interventions: Drug: phosphatidylcholine-curcumin complex supplement
- Placebo curcumin capsules (Placebo Comparator): Dose will be matching placebo capsules daily, orally for 24 weeks
  Interventions: Drug: Placebo curcumin capsule

INTERVENTIONS:
Drug: phosphatidylcholine-curcumin complex supplement — a dietary curcumin supplement given at two different doses
  Other Names: Meriva®
  Arms: Curcumin 1000mg capsules; Curcumin 500mg capsules
Drug: Placebo curcumin capsule — matching placebo to active curcumin capsules
  Arms: Placebo curcumin capsules

SUMMARY:
This is a single-center, randomized, double-blinded, placebo-controlled, parallel treatment groups phase 2a study of curcumin for pediatric nonalcoholic fatty liver disease (NAFLD).

DETAILED DESCRIPTION:
30 subjects ages 8-17y, with biopsy-proven NASH/NAFLD (≤ 730 days prior to registration and a NAFLD Activity Score (NAS) of ≥3) and serum ALT at screening ≥ 50 IU/L at enrollment. Eligible participants will receive curcumin 500 mg, 1.0 g or placebo for 24 weeks, randomized 1:1:1. The primary outcome of the study will determine whether 24 weeks of curcumin supplementation compared to matching placebo improves measures of nonalcoholic fatty liver disease (NAFLD) as determined by relative improvement in serum ALT from baseline. The hypothesis is that curcumin will significantly decrease ALT relative to placebo in children with NAFLD.

ELIGIBILITY:
Inclusion Criteria:

* Age 8-17 years at initial screening interview
* Histological evidence of NAFLD with or without fibrosis and a NAFLD activity score (NAS) of ≥3, on a liver biopsy obtained no more than 730 days prior to enrollment
* Serum ALT at screening ≥ 50 IU/L

Exclusion Criteria:

* Significant alcohol consumption or inability to reliably quantify alcohol intake
* Use of drugs historically associated with NAFLD (amiodarone, methotrexate, systemic glucocorticoids, tetracyclines, tamoxifen, estrogens at doses greater than those used for hormone replacement, anabolic steroids, valproic acid, other known hepatotoxins) for more than 2 consecutive weeks in the past year prior to randomization
* New treatment with vitamin E or metformin started in the past 90 days or plans to alter the dose or stop over the next the 24 weeks. A stable dose is acceptable.
* Prior or planned bariatric surgery
* Uncontrolled diabetes (HbA1c 9.5% or higher within 30 days prior to enrollment)
* Presence of cirrhosis on liver biopsy
* Stage 2 Hypertension or >140 systolic or >90 diastolic at screening
* Current daily use of nonsteroidal anti-inflammatory drugs (NSAIDs)
* Platelet counts below 100,000 /mm3
* Clinical evidence of hepatic decompensation (serum albumin < 3.2 g/dL, international normalized ratio (INR) >1.3, direct bilirubin >1.3 mg/dL, history of esophageal varices, ascites, or hepatic encephalopathy)
* Evidence of chronic liver disease other than NAFLD:

  * Biopsy consistent with histological evidence of autoimmune hepatitis
  * Serum hepatitis B surface antigen (HBsAg) positive.
  * Serum hepatitis C antibody (anti-HCV) positive.
  * Iron/total iron binding capacity (TIBC) ratio (transferrin saturation) > 45% with histological evidence of iron overload
  * Alpha-1-antitrypsin (A1AT) phenotype/genotype ZZ or SZ
  * Wilson's disease
* History of biliary diversion
* History of kidney disease and/or estimated glomerular filtration rate (eGFR) < than 60 mL/min/1.73 m2 using Schwartz Bedside GFR Calculator for Children isotope dilution mass spectroscopy (IDMS)-traceable
* Known Human Immunodeficiency Virus (HIV) infection
* Active, serious medical disease with life expectancy less than 5 years
* Active substance abuse including inhaled or injected drugs, in the year prior to screening
* Pregnancy, planned pregnancy, potential for pregnancy and unwillingness to use effective birth control during the trial, breast feeding
* Participation in any clinical/investigational trial within the prior 150 days and during the study.
* Any other condition which, in the opinion of the investigator, would impede compliance or hinder completion of the study
* Inability to swallow capsules
* Known allergy to curcumin or any of its components
* Failure of parent or legal guardian to give informed consent or subject to give informed assent

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2019-12-09 (Actual); Primary Completion 2020-04-22 (Actual); Study Completion 2020-04-22 (Actual)

PRIMARY OUTCOMES:
Change in serum alanine aminotransferase (ALT) from baseline. | 24 weeks
  ALT value in U/L

SECONDARY OUTCOMES:
Relative change in ALT compared to baseline ALT | 24 weeks
  ALT value in U/L
Proportion of patients achieving normalization of ALT | 24 weeks
  ALT value in U/L
Change in serum aspartate aminotransferase (AST) | 24 weeks
  AST value in U/L
Change in serum gamma-glutamyl transpeptidase (GGT) | 24 weeks
  GGT value in U/L
Change in ALT at 12 weeks compared to baseline ALT | 12 weeks
  ALT value in U/L
Change in Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) compared to baseline | 24 weeks
  is an equation which indicates the degree of insulin resistance, where higher scores equate to greater insulin resistance. HOMA-IR is calculated as fasting (Glucose (mmol/L) x insulin (pmol/L))/22.5. A HOMA-IR value >2.0 in prepubertal children and >2.6 in pubertal children, may be considered a warning sign for pediatricians to further investigate insulin resistance
Change in Weight | 24 weeks
  kilograms (kg)
Change in Waist circumference | 24 weeks
  centimeters (cm)
Change in Waist to Hip ratio | 24 weeks
  ratio of the circumference of the waist to that of the hips. This is calculated as waist measurement divided by hip measurement (W ÷ H).
Change in Body-mass Index Z- Score | 24 weeks
  Body mass index z-scores is calculated using age, gender, height and weight and calculated using 2000 CDC Growth Charts for norms.
Change in serum lipids compared to baseline | 24 weeks
  lipid profiles
Change in High Sensitivity C-Reactive Protein (hsCRP) compared to baseline | 24 weeks
  serum marker of inflammation (mg/L)
Change in Pediatric Quality of Life Inventory (PedsQL) Score scores compared to baseline | 24 weeks
  Pediatric Quality of Life Inventory (PedsQL) version 4.0 is completed by both the child and parent/caregiver, and is composed of 23 items comprising 4 dimensions: Physical Functioning, Emotional Functioning, Social Functioning, and School Functioning. Scores are transformed on a scale from 0 to 100, with higher scores indicating better health-related quality of life. Physical Health Summary Score =Physical Functioning Scale Score. Psychosocial Health Summary Score = Sum of items over the number of items answered in the Emotional, Social, and School Functioning Scales.
Change in Intrahepatic fat content and liver stiffness | 24 weeks
  Hepatic fat content and liver stiffness will be measured by CAP and VCTE (Fibroscan®)
Change in frequency of adverse events compared to baseline | 24 weeks
  Numbers of adverse events reported

OTHER OUTCOMES:
Plasma concentrations of curcumin and active metabolites from baseline to 24 weeks. | Day 0 pre-dose and 1, 2, 4, 6, 8 hours post-dose; Day 14; Day 28; Day 84 and Day 168
  Pharmacokinetic analysis
Change in interleukin 6 (IL-6) | 24 weeks
  cytokine protein involved in the pro-inflammatory and anti-inflammatory response
Change in interleukin 8 (IL-8) | 24 weeks
  cytokine protein involved in the pro-inflammatory and anti-inflammatory response
Change in (TNF-a) Tumor Necrosis Factor alpha | 24 weeks
  cytokine protein involved in the pro-inflammatory and anti-inflammatory response
Change in Plasminogen Activator Inhibitor (PAI-1) | 24 weeks
  cytokine protein involved in the pro-inflammatory and anti-inflammatory response
Change in adiponectin | 24 weeks
  cytokine protein involved in the pro-inflammatory and anti-inflammatory response

CONTACTS AND LOCATIONS:
Overall Officials: Joel E Lavine, MD, PhD, Principal Investigator — Columbia University

IPD SHARING:
Plan to Share IPD: No